CLINICAL TRIAL: NCT02562261
Title: Platelet Reactivity During Different Stages of Sepsis
Brief Title: Platelet REactivity in Sepsis Syndrome (PRESS)
Acronym: PRESS
Status: Completed | Type: Observational
Sponsor: Charalambos .A. Gogos (Other)
Collaborators: Hellenic Society for Chemotherapy : Hellenic Sepsis Study Group (Unknown); University Hospital of Patras (Other)
Responsible Party: Sponsor-Investigator, Charalambos .A. Gogos, Professor in Internal Medicine and Infectious Diseases, University Hospital of Patras
Organization: University Hospital of Patras (Other)
Other Study IDs: 24958/19-12-13
Record Dates: First submitted 2015-09-15; First posted 2015-09-29 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Sepsis Syndrome
Keywords: sepsis; platelet; platelet reactivity; P2Y12
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Healthy
- Uncomplicated Infection: Showing signs of infection as defined by International Sepsis Definitions Conference 2003
- Sepsis: Sepsis is defined as systemic inflammatory response syndrome (i.e. presence of two or more of the following
  1. Temperature of <36 °C (96.8 °F) or >38 °C (100.4 °F)
  2. Heart rate >90bpm
  3. Respiratory rate >20/min or PaCO2<32 mmHg (4.3 kPa)
  4. WBC <4x109/L (<4000/mm³), >12x109/L (>12,000/mm³), or 10% bands in response to an infectious process..
- Severe Sepsis/Septic Shock: Severe sepsis is defined as sepsis with sepsis-induced organ dysfunction or tissue hypoperfusion [manifesting as hypotension, elevated lactate (serum lactate 2 times the upper limit of normal), or decreased urine output (urine output < 0.5 ml/kg/hr)] Septic shock is defined as severe sepsis plus persistently low blood pressure (< 5th percentile for age or systolic blood pressure < 2 standard deviations below normal for age) following the administration of intravenous fluids.

SUMMARY:
Activation of blood platelets is a typical finding in patients with systemic inflammation and sepsis.They seem to mediate key pro-inflammatory mediator secretion, immune-cell activation while their adhesion to the endothelium enhances the pro-coagulatory activity of endothelial cells impairing microcirculation thus, may lead to multiple organ dysfunction. However, the exact effects of bacterial products on platelet function have not been found to be consistent and may vary according to the species, the timing of the study, and the pathogenesis of sepsis. Data vary, including both increased and decreased platelet reactivity and aggregation among patients with sepsis compared to healthy controls. Defining platelet's behaviour during sepsis is particularly important in view of recent findings revealing potential association between antiplatelet therapy and reduction in short term mortality, incidence of acute lung injury and intensive care unit admission in critically ill patients.This study aims to measure P2Y12 mediated platelet reactivity, -using the point-of-care P2Y12 VerifyNow assay, in platelet reactivity units (PRU)- along different stages of sepsis, including bacteremia/uncomplicated infection, sepsis, severe sepsis and septic shock. Subgroup follow up of patients going along different stages will also be performed. At the end of this study analysis of clinical and laboratory findings in correlation with platelet reactivity will be performed to assess platelet aggregation during sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting 0-8 hours post admission with signs of one of the following i) uncomplicated infection/bacteremia ii) sepsis iii) severe sepsis iv) septic shock
* 30 healthy subjects
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Inability to give informed consent
* PLTs<70.000/ul or PLTs>741.000 ul
* Ht<25% or Ht>52%
* History of P2Y12 or GPIIb/IIIainhibitors the last 15 days prior assortment
* Patients with inherited (vonWillebrand factor deficiency, Glanzmann thrombasthenia, Bernard-Sulier syndrome) or established acquired platelet disorders (HIT)
* Patients undergoing hemodialysis
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 3 months.
* Previous history of immunologic disease (neoplasm, autoimmune disorders, HIV)
* Subjects receiving daily treatment with immune-modulating regimens.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Within 0-8 hours of presentation in emergency department patients will be assessed and assigned upon their health status in four distinct groups of uncomplicated infection/bacteraemia , sepsis, severe sepsis/septic shock as this is defined by International Sepsis Definitions Conference. Thirty five healthy volunteers will serve as a control group.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
P2Y12 mediated Platelet Reactivity on presentation | 0 hours post presentation
  Measurement of P2Y12 mediated platelet reactivity of patients in different study groups i.e healthy controls, uncomplicated infection, sepsis, severe sepsis/septic shock in P2Y12 reactivity units (PRU). PRU measurement will take place on time of presentation and recognition of signs of infection
Comparison of P2Y12 mediated Platelet Reactivity between study groups | at 1 year
  Measurements of P2Y12 mediated platelet reactivity of different study groups that have taken place on presentation will be compared following completion of study recruitment

SECONDARY OUTCOMES:
Serum levels of pro-inflammatory mediators in various study groups | 1 month to 1 year
  Patient serum will be collected and cytokines will be measured in all patients
Correlation between serum levels of pro-inflammatory mediators and measured PRU between various study groups | 1 month to 1 year
  Following measurement of serum cytokines (outcome 3), assessment of potential correlation with PRU will be performed
Repeated measurement of PRU in the same subject when transiting from one group to another | 1 hour to 1 month
  Patients transiting from one stage of sepsis to another (for example severe sepsis to healthy state OR from uncomplicated infection to sepsis) will be repetitively measured to assess platelet reactivity alteration

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Gogos, MD,PhD, Study Director — University Hospital of Patras; Karolina Akinosoglou, MD,PhD, Principal Investigator — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

REFERENCES:
- See also: Platelet reactivity in sepsis syndrome: results from the PRESS study — https://www.ncbi.nlm.nih.gov/pubmed/28840345